CLINICAL TRIAL: NCT07310953
Title: Clinical Utility of the Numerical Verbal Scale (NVS) and the Pain and Functional Activity Scale (PFAS) in the Management of Rescue Analgesia in Acute Postoperative Pain. Randomized Study.
Acronym: EVN/EDAF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EVN/EDAF; 2025/306 (Other: Galician Ethics Committee for Medicinal Products (CEIm-G))
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-10

CONDITIONS: Analgesia; Post Operative Pain; Acute Pain; Functional; Anesthesia
Keywords: numerical verbal scale; Functional Activity Score
MeSH Terms: conditions — Agnosia; Pain, Postoperative; Acute Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single blind for the data analyzer in which the patients of the scheduled surgeries selected in the selection criteria will be included.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Rescue analgesia if EVN>4
  Interventions: Procedure: Group A: Rescue analgesia if NVS>4
- Group B (Experimental): Rescue analgesia if EVNm >4 + FAS C
  Interventions: Procedure: Group B: Rescue analgesia if NVSm > 4 + FAS C

INTERVENTIONS:
Procedure: Group A: Rescue analgesia if NVS>4 — Rescue analgesia will be self-administered by the patient, when post-surgical pain is moderate to severe, using morphine PCA at a dose of 0.075 mg/kg maximum every 15 minutes, up to a maximum of 3 times per hour, provided they meet the criteria described for the group to which they have been assigned.
  Arms: Group A
Procedure: Group B: Rescue analgesia if NVSm > 4 + FAS C — Rescue analgesia will be self-administered by the patient, when post-surgical pain is moderate to severe and this pain interferes with and limits functional activity, using morphine PCA at a dose of 0.075 mg/kg maximum every 15 minutes, up to a maximum of 3 times per hour, provided they meet the criteria described for the group to which they have been assigned.
  Arms: Group B

SUMMARY:
Adequate postoperative pain management, along with mobilization and early oral nutrition, is the foundation for optimal recovery after surgery.

Unidimensional pain scales (Numerical Verbal Rating Scale - NRS, Visual Analogue Scale - VAS, Categorical Scale - CRS, Facial Pain Scale - FPS) do not adequately reflect a patient's actual analgesic needs. Basing analgesic treatment on the classic algorithm of administering opioids if pain is greater than 4 on the NRS, without considering functional impairment, has been shown to be a cause of overtreatment in surgical wards.

The Functional Activity Score (FAS) is the simplest scale, designed for bedside application and geared toward therapeutic decision-making. R: Able to perform any activity; B: Pain prevents some activity; C: Unable to perform any activity.

Given the need to standardize functional limitation when measuring postoperative pain, we propose the Pain and Functional Activity Scale (PFAS), which combines the NVA (Non-Visual Analogue Scale) with the Functional Activity Scale. Specifically, pain on movement would be recorded using the NVA in motion (NVAm), along with functional limitation (A, B, or C). The rescue analgesia treatment algorithm adapted to the PFAS would involve treating patients with pain greater than 4 on the NVA whenever it represents a severe limitation of their functional activity (C).

In this study, we aim to evaluate whether there are significant differences in the proportion of patients who meet the criteria for needing rescue analgesia according to the NVA compared to the proportion of patients who meet the criteria for needing rescue analgesia established by the PFAS, during the 2-day postoperative period.

To this end, an experimental, longitudinal, prospective, randomized, single-blind study for the data analyzer will be carried out, where a group that will receive rescue analgesia if VNS>4 and another if VNSm>4 + FAS C will be compared in the first two days of postoperative surgical patients of the surgeries selected in the EOXI of Vigo.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled surgery with VATS admission
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Cognitive-mental deficit assessed using the Pfeiffer questionnaire. Patients with more than two errors if they have a university degree and more than three errors if they do not have a university degree are excluded from the study.
* Allergy to any of the analgesic drugs listed on the data collection sheet (Paracetamol / NSAIDs / Metamizole / Dexamethasone / Local anesthetics / Morphine / Fentanyl).
* Patients who, in the preoperative survey, present any degree of functional limitation according to the FAS scale (Grade B and C).

Withdrawal Criteria:

* If the patient withdraws consent.
* If the patient experiences delirium, as measured by a positive CAM (Confusion Assessment Method) scale, following surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
NVS | Day 0 (before the surgical intervention), at 24 and 48 hours and in case rescue analgesia is requested.
  Resting Numerical Verbal Scale (NVS), indicate one of the following options (0 = no pain 10 = the worst pain imaginable): 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10.
mNVS | Day 0 (before the surgical intervention), at 24 and 48 hours and in case rescue analgesia is requested.
  Moving Numerical Verbal Scale (mNVS), indicate one of the following options (0 = no pain 10 = the worst pain imaginable): 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10.
FAS | Day 0 (before the surgical intervention), at 24 and 48 hours and in case rescue analgesia is requested.
  Functional Activity Score (FAS): After evaluating the following activities: Sitting, Walking, Rehabilitation, Respiratory Physiotherapy; indicate how pain interferes with your functional activity and rank them from best to worst:
  * A: Able to perform any activity (performs all 4 activities without limitation)
  * B: Pain prevents some activity (unable to perform between 1 and 3 of the activities)
  * C: Unable to perform any activity (is unable to perform any of the activities)

SECONDARY OUTCOMES:
Age | Day 0 (before the surgical intervention)
  Patient age in years
Gender | Day 0 (before the surgical intervention)
  Patient gender (Female, Male)
BMI | Day 0 (before the surgical intervention)
  Patient body mass index
Pfeiffer | Day 0 (before the surgical intervention)
  Cognitive-mental deficit assessed according to the Pfeiffer questionnaire:
  1. What is today's date (day, month, year)? 2. What day of the week is it today? 3. Where are we now (place or building)? 4. What is your telephone number? (or your address if you don't have a telephone) 5. How old are you? 6. What is your birth year? 7. Who is the current Prime Minister? 8. Who was the previous Prime Minister? 9. What is your mother's second surname? 10. Subtract 3 each time from the number 20.
  Patients with more than 2 errors if they have a university degree and more than 3 errors if they do not have a university degree will be excluded from the study.
  After completing the questionnaire, the variable is recorded as yes/no.
ASA | Day 0 (before the surgical intervention)
  Anesthetic risk scale (ASA), indicate one of the following options: 0-No risk, 1-Low risk, 2-Moderate risk, 3-High risk
Risk factors associated with persistent postoperative pain | Day 0 (before the surgical intervention)
  Risk factors associated with persistent postoperative pain, indicate the following option(s):
  * Treatment with antidepressants
  * Treatment with anxiolytics/benzodiazepines
  * Catastrophizing (Yes: moderate-to-high risk/ No: low risk) [The Pain Catastrophizing Scale - abbreviated PCS-4 - will be applied). (4-8 low risk; 9-12 moderate risk; 13-16 high risk)
  * Chronic preoperative pain [NV >4 for more than 3 months, in any location]
  * Use of strong opioids and/or tramadol at doses greater than 60 mg/day for more than 3 months
  * History of use of opiates, cannabis, lysergic acid diethylamide (LSD), 3,4-methylenedioxymethamphetamine (MDMA)
  * History of alcohol consumption >40 grams/day in men and >20 grams/day in women
Procedure | Day 1 (after the surgical intervention)
  Surgical procedure, indicate one of the following options: Upper lobectomy, Middle lobectomy, Lower lobectomy.
Surgery location | Day 1 (after the surgical intervention)
  Surgery location, indicate one of the following options: Right, Left.
Anesthetic technique | Day 1 (after the surgical intervention)
  Anesthetic technique, indicate one of the following options: Inhalational general anesthesia, Intravenous general anesthesia
Intraoperative analgesia guidelines | Day 1 (after the surgical intervention)
  Intraoperative analgesia guidelines, choose the type of drug: Fentanyl, paracetamol, NSAIDs
Confusión Assessment Method (CAM) | at 24 and 48 hours
  Postoperative Neurological Status of the Patient by Confusión Assessment Method:
  1. Acute Onset and Fluctuating Course
  2. Inattention
  3. Disorganized Thinking
  4. Altered Level of Consciousness
  1. Alert (normal) 2. Vigilant (hyperalert, very sensitive to environmental stimuli) 3. Lethargic (inhibited, drowsy) 4. Stuporous (difficult to awaken)
  For a diagnosis of delirium, the first two criteria and at least one of the last two are necessary.
  After completing the questionnaire, the variable is recorded as yes/no.
Analgesia guidelines in the post-surgical intensive care unit | at 24 and 48 hours
  Analgesia guidelines in the post-surgical intensive care unit, indicate
  * Rescue dose of morphine (PCA)
  * Total dose in mg
Side effects of analgesia | at 24 and 48 hours
  Side effects of analgesia, indicate from the following options:
  * Nausea / Vomiting
  * Postoperative ileus [Oral intolerance and/or need for nasogastric tube]
  * Mental confusion / Hallucinations
  * Sedation [Ramsey Scale] see appendix.
  * Pruritus
  * Respiratory depression [Respiratory rate < 12 breaths/min, requiring therapeutic maneuvers]
  * Other (specify)
Nighttime rest | at 24 and 48 hours
  Nighttime rest at 24 and 48 hours: Sleep scale. To answer the question "How do I sleep?" the patient responds on a scale from 0 (I don't sleep at all) to 10 (I sleep perfectly).
Desire for more analgesia | at 48 hours
  Desire for more pain relief than received (Yes, No, Don't know)
Satisfaction with pain management therapy | at 48 hours
  Satisfaction with pain management therapy using 4 categories:
  * Very dissatisfied
  * Dissatisfied
  * Satisfied
  * Very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Álvaro Cunqueiro, Vigo, Spain

IPD SHARING:
Plan to Share IPD: No